CLINICAL TRIAL: NCT02380183
Title: A Randomized Controlled Study Comparing Needle-Guided vs Free-Hand Technique in Performing Brachial Plexus Blockade
Brief Title: Needle-Guided vs Free-Hand Technique in Performing Brachial Plexus Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: CIVCO Medical Solutions (Unknown)
Responsible Party: Principal Investigator, Amaresh Vydynathan, Assoc. Prof. Anesthesiology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-3414
Record Dates: First submitted 2015-01-30; First posted 2015-03-05 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Needle Guidance; Nerve Blocks
Keywords: anesthesia; nerve block; needle guidance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): Civco needle guidance device will be used while the nerve block is performed.
  Interventions: Device: Civco Needle Guidance Device
- Standard of Care (No Intervention): Needle guidance device will not be used while nerve block is performed; nerve block is performed by hand alone.

INTERVENTIONS:
Device: Civco Needle Guidance Device — Needle guidance device will be used while nerve block is performed.
  Arms: Intervention

SUMMARY:
This is an openly randomized controlled parallel group study evaluating the effectiveness of using a guided approach and free-hand approach in performing upper extremity regional blocks. Potential subjects for this study are the patients who are scheduled for upper extremity surgeries requiring supraclavicular and interscalene brachial plexus blocks at Montefiore Medical Center.

Rotating residents who are participating in the study will be randomly assigned either to perform block under guided approach (with the help of needle guidance) or free-hand without the needle guidance. All the blocks will be single injection blocks utilizing the in-plane technique for needle insertion which is the usual protocol in our institution. Each resident will be performing one interscalene block with the device and one without the device and one supraclavicular block with device and one without the device. An independent observer will be present during the case and will be responsible for recording the time taken to perform the block, number of times the needle has been redirected and the number of times the needle is reinserted. This observer will also administer the satisfaction questionnaire. Number of time needle is redirected and number of times reinserted is also a self reported assessment by the physician who is performing the block. Efficacy of the block will be assessed by the standard of care practiced at our center.

DETAILED DESCRIPTION:
Objectives

1. The primary end point of the study is to evaluate the time taken to complete blocks with and without the use of the needle guidance device. (Start time is considered as the first skin touch by the needle until the completion of the block. Completion of the block is defined as withdrawing the needle completely out of the body). The principal investigator/co-investigator and an independent observer will be recording the time taken to complete the block.
2. Ease of the technique- (Will be assessed with a short questionnaire survey at the end of the procedure). Immediately after the block is finished, the performing physician will be requested to fill out the questionnaire.
3. Number of times needle needs to be re-directed. This is self a reported measurement. The person performing the block, investigators (attending physician) and an independent observer will be recording number of times the needle was manipulated.
4. Number of times needle was pulled out entirely out of the body and reinserted. This is also a self reported measurement.
5. Efficacy of the blocks performed will be assessed (This is part of the routine standard of care assessing the blocks.)
6. Total amount of time taken to complete the whole procedure (Starting from the first time the ultrasound probe was placed on the patient to the withdrawal of the needle after completing the procedure)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* ASA 1-3 for upper extremity surgery receiving interscalene or supraclavicular blockade
* Able to understand and sign the informed consent

Exclusion Criteria:

* Patient refusal of regional anesthesia
* Any contraindications to regional anesthesia
* Any anatomical or neurological disorders (also applicable to the diagnosis made by the anesthesiologist prior to randomization of the patient)
* Any other condition /diagnosis by the anesthesiologist that could compromise performing the block

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amaresh Vydyanathan, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Full Range); unit: years] | 56 [41 to 71] | 50 [34 to 66] | 53 [34 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 18 | 14 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Needle Time;
Description: needle insertion to needle withdrawal
Time Frame: Needle insertion to needle withdrawal, up to 20 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 36 | 34
seconds | 106 [92 to 162] | 197 [140 to 278]

2. Secondary Outcome: Nerve Block Procedure Time
Description: How long the procedure takes in minutes, starting from ultrasound contact with skin to needle withdrawal.
Time Frame: time from ultrasound contact with skin to needle withdrawal, up to 20 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 36 | 34
seconds | 86 [76 to 146] | 126 [94 to 126]

ADVERSE EVENTS:
Time Frame: There were no adverse events reported throughout the duration of our study.
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
A limitation of this study was that most of the clinicians using the device were either senior residents (CA-3's), or fellows. It is possible that this device could provide more or less benefit in newer trainees.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No